CLINICAL TRIAL: NCT01463254
Title: A Prospective Observational Study of the Clinical Performance of Femplant in Pakistan
Status: Completed | Type: Observational
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 10231
Record Dates: First submitted 2011-10-13; First posted 2011-11-01 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Contraception
Keywords: Femplant; AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU international units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surveillance: - a surveillance cohort of 300 women who will report back to the clinic during 12 months after enrolment only if they have complications, medical problems, pregnancy, or want to remove the implant
- Prospective: a prospective cohort consisting of 300 women who will be followed-up 3 and 12 months after enrollment

SUMMARY:
This will be a non-comparative prospective observational study of women using Femplant as a primary method of contraception in Pakistan.

DETAILED DESCRIPTION:
This will be a non-comparative prospective observational study of women using Femplant as a primary method of contraception in Pakistan. It will be conducted in close collaboration with the Pakistan MoH and Marie Stopes Society, Pakistan in several MoH-affiliated and Marie Stopes Society clinics that have experience with implants and sufficient expected flow of implant users per month. We will enroll a total of 600 women divided into two cohorts in this one-year prospective study:

* a prospective cohort consisting of 300 women who will be followed-up 3 and 12 months after enrolment; and
* a surveillance cohort of 300 women who will report back to the clinic during 12 months after enrolment only if they have complications, medical problems, pregnancy, or want to remove the implant

The main study outcomes are pregnancy, immediate and delayed complications associated with insertion or removal, adverse events, early discontinuation and reasons for discontinuation, and level of women's satisfaction with Femplant services.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion, a woman must:

  * be aged 18-44 years, inclusive
  * be willing to sign an informed consent document
  * agree to return for follow-up visits
  * have decided to receive Femplant as a method of contraception and met the clinic criteria for eligibility of this method of contraception

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women using Femplant as a primary method of contraception in Pakistan
Sampling Method: Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
pregnancy | 12 months
  measure number of pregnancies while using implant
Immediate and Delayed Complications | 12 months
  Measure Immediate and delayed complications associated with insertion or removal of implant
Adverse events | 12 months
  to record any adverse events associated with the implant
Measure number of participants who discontinue from the study | 12 months
  Measure number of participants who discontinue from the study and the reasons for discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Paul Feldblum, PhD, Study Director — FHI 360; Syed Khurram Azmat, MD, Principal Investigator — Marie Stopes Society, Pakistan; Adrienne Testa, Study Chair — Marie Stopes Internatioanl
Locations (1):
- Marie Stopes Society clinics, Pakistan, Pakistan, Pakistan